CLINICAL TRIAL: NCT00700466
Title: Beta-adrenoceptor Blockade Prior to Induction of Anesthesia for Improvement of Depressed Autonomic Regulation
Brief Title: Intravenous Beta-blockade for Improvement of Autonomic Activity
Status: Completed | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Jens Scholz, Chair of the Department of Anaesthesiology and Intensive Care Medicine, University Hospital Schleswig-Holstein, Campus Kiel, Germany
Other Study IDs: Hanss_EA 162/07
Record Dates: First submitted 2008-06-13; First posted 2008-06-18 (Estimated); Last update posted 2010-01-18 (Estimated); Status verified 2009-02

CONDITIONS: Hypertension; Tachycardia; Heart Rate Variability
Keywords: Outcome assessment, patients;; autonomic nervous system;; perioperative care;; adrenergic beta antagonist; Autonomic regulation; Perioperative beta-blockade; outcome
MeSH Terms: conditions — Hypertension; Tachycardia | interventions — Metoprolol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Patients with hypertension and/or tachycardia prior to induction of anesthesia requiring i.v. beta-blockade for treatment of raised hemodynamic
  Interventions: Drug: i.v. beta-blocker infusion (metoprolol)
- 2: Patients with normal hemodynamic values prior to induction of anesthesia not requiring treatment

INTERVENTIONS:
Drug: i.v. beta-blocker infusion (metoprolol) — A beta-blocker (metoprolol) will be infused for treatment of hypertension and/or tachycardia prior to induction of anesthesia aiming at decrease of blood pressure and heart rate to normal limits
  Other Names: Metorpolol, Lopresor(R)
  Groups: 1

SUMMARY:
Chronic beta-adrenoceptor blockade is known to improve outcome of high risk patients whereas amelioration of autonomic activity was demonstrated to be a major cause of outcome improvement. Therefore, perioperative beta-adrenoceptor blockade is recommended in patients with Revised Cardiac Risk Index score of three or greater. The investigators hypothesise that preoperative intravenous beta-adrenoceptor blockade for treatment of hypertension and/or tachycardia improves autonomic activity reflected by increase of Total Power of Heart Rate Variability.

Material and Methods: After IRB approval 20 patients scheduled for elective cardiac surgery were included into the study. Routine medication was continued throughout the study as recommended by the guidelines. HRV (TP and Low to High Frequency ratio (LF/HF) reflecting sympathetic to parasympathetic balance) was analysed prior to induction of general anesthesia and beta-adrenoceptor blockade in all patients (Baseline). Patients were assigned by their baseline hemodynamics. Patients with hypertension (systolic blood pressure > 140mmHg or diastolic blood pressure > 90mmHg) or tachycardia (heart rate > 80bpm) were assigned to group BETA-BLOCK. In this group metoprolol-boli (2mg) were administered intravenously in stepwise manner until hemodynamic values decreased to normal. Total dosage was recorded. After normalisation of hemodynamics, second HRV analysis was performed (Intervention). Normotensive and normocardic patients were assigned to group CONTROL. No intervention was performed. Statistics: Mann Whitney U test for comparison between groups and between events Baseline and Intervention within group BETA-BLOCK, p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for coronary artery bypass surgery
* Ejection fraction > 30 %
* Informed consent

Exclusion Criteria:

* Emergency cases
* Myocardiac infraction within 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for coronary artery bypass surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-03 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Improvement of heart rate variability reflecting autonomic activity in the course of i.v. beta-blockade | Baseline, after i.v. beta-blockade, 6 months after discharge

SECONDARY OUTCOMES:
Hospital stay, one-year cardiac mortality and morbidity after discharge | Postoperatively until discharge, between discharge and 1 year after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hanss, MD, Principal Investigator — Consultant in Anesthesiology, Dep. of Anesthesiology and Intenisve Care Medicine, University Hospital Schleswig-Holstein, Campus Kiel, Germany
Locations (1):
- University Hospital Schleswig-Holstein, Campus Kiel, Germany, Kiel, Schleswig-Holstein, Germany